CLINICAL TRIAL: NCT02073214
Title: Effects of Oral Probiotic Supplementation on the Clinical Status of Very-low-birth-weight Preterm Neonates. Multi-centre, Randomised, Double-blind, Placebo-controlled Clinical Study.
Brief Title: Effects of Oral Probiotic Supplementation on the Clinical Status of Very-low-birth-weight Preterm Neonates.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IBSS Biomed S.A. (Industry)
Collaborators: Ministry of Science and Higher Education, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PB-DM/SBK-NEC-01/11
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Late Onset Neonatal Sepsis; Necrotizing Enterocolitis; Infant, Very Low Birth Weight
MeSH Terms: conditions — Neonatal Sepsis; Enterocolitis, Necrotizing | interventions — Probiotics; Food

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Experimental): Single dose of probiotic, was administered enterally twice daily with food (in the morning and in the evening). The first dose of probiotic was administered within the first 48 hours after birth. The probiotic administration was continued for 6 weeks or until hospital discharge (whichever was earlier).
  Discontinuation of the enteral nutrition was equivalent with discontinuation of the administration of the probiotic. If the probiotic was discontinued for more than 7 days, the patient was withdrawn from the study.
  Interventions: Other: Probiotic
- Placebo (Placebo Comparator): Single dose of placebo was administered enterally twice daily with food (in the morning and in the evening). The first dose of placebo was administered within the first 48 hours after birth. The placebo administration was continued for 6 weeks or until hospital discharge (whichever was earlier).
  Discontinuation of the enteral nutrition was equivalent with discontinuation of the administration of the placebo. If the placebo was discontinued for more than 7 days, the patient was withdrawn from the study.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Probiotic — Standard treatment plus probiotic
  Other Names: Food for special medical purposes
  Arms: Probiotic
Other: Placebo — Standard treatment plus placebo
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the safety of a probiotic foodstuff and its influence on emergence and development of natural intestinal flora and the clinical status of premature very low birth weight neonates. The study was also intended to investigate reduction of colonisation by pathogenic bacteria and to estimate the incidence of gastrointestinal disorders.

Probotic bacteria contained in the investigational product administered directly after birth are beneficial for the development of normal gut microflora and can prevent or significantly limit gastrointestinal colonisation by pathogenic bacteria and the development of pathogenic flora in a hospital setting. Permanent colonisation with commensal flora in very early life improves gastrointestinal function in premature neonates by reducing the onset of or by decreasing the severity of the signs and symptoms of feeding intolerance and generalised bacterial infections, including sepsis and necrotizing enterocolitis.

DETAILED DESCRIPTION:
Neonates defined as having very low birth weight (VLBW) are found to have a number of conditions typical for this period of life and body weight at birth. Perinatal and neonatal infections are relatively common in these babies, which can be attributed to their immunological immaturity (immature cellular or humoral immune responsiveness) and insufficient gastrointestinal tract colonisation by non-pathogenic bacteria, the presence of which depends on the type of delivery, feeding and environment in which the neonates are nursed.

Neonates admitted to neonatal intensive care units, particularly low birth-weight neonates born prematurely or with congenital disorders, are most susceptible. Probiotics administered to neonates are known to compete with pathogenic bacteria for essential nutrients and receptor sites, and to enzymatically modify toxin receptors. They are also known to produce antimicrobial substances, acidify the intestinal environment and stimulate the immune system, helping it reach full maturity. These are the reasons why intestinal microflora normalisation with the help of probiotics can be beneficial for VLBW neonates, especially those requiring intensive medical care.

In a review of clinical studies on the use of probiotics in NEC prevention in neonates, demonstrated beneficial effects of probiotics in a group of VLBW neonates compared to placebo. There are scientific reasons to believe that probiotics administered to neonates modulate the composition of the gut flora colonising the intestinal tract and are beneficial for the development and maturity of the immune system. In hitherto clinical studies, specific probiotic strains were found to provide beneficial effects by limiting infections in the neonatal period, including necrotizing enterocolitis in VLBW neonates.

The purpose of this multicentre, randomized study was to investigate whether the use of a probiotic preparation containing Lactobacillus rhamnosus KL53A and Bifidobacterium breve PB04 influence on emergence and development of natural intestinal flora and the clinical status of premature very low birth weight neonates and reduction of colonisation by pathogenic bacteria and to estimate the incidence of gastrointestinal disorders. The study took place between April 2012 and July 2013 in eight study centres in Poland. It was conducted in accordance with the original protocol and according to ICH-GCP requirements.

The duration of subject's participation in the trial was approximately 49 days, or until they were withdrawn or discharged from the hospital, whichever came earlier, prior to day 49.

As the trial did not concern medicinal product but the foodstuff (food for special medical purpose) it did not require Authority approval but was only subject to relevant Ethics Committee approval.

The study only included neonates who fulfilled the eligibility criteria, after obtaining an informed consent from their parents/legal guardians, to have their baby enrolled in the study and randomized into one of the two study groups: probiotic or placebo. Investigational product were administered during the first 48h of life, at the time of the enteral feed.

Efficacy evaluation was to determine whether the investigational product positively influences the emergence and progressive development of the natural gut flora and the clinical status of preterm VLBW neonates. As part of the efficacy evaluation, it was also examined whether the probiotic agent has the capacity to inhibit pathogenic colonisation and to reduce the incidence of gastrointestinal disorders, as compared to placebo.

Safety was evaluated by determining whether investigational product in VLBW preterm neonates increases AE/SAE incidence and influences the type of adverse events and serious adverse events as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Infants ≥ 750 g and ≤ 1800 g at birth
2. Gestational age of ≤ 34 weeks
3. Mother's age ≥ 18 years
4. Possibility of feeding by enteral route
5. Possibility of enrolment ≤ 48 hours of age
6. Caucasian race
7. Parent-legal guardian informed consent obtained in writing

Exclusion Criteria:

1. Infants < 750 g and > 1800 g at birth
2. Gestational age of > 34 weeks
3. Mother's age < 18 years
4. Contraindicated to enteral nutrition within the first 48 hours of life
5. Birth asphyxia (Apgar score: 0-3)
6. Major congenital abnormalities, including gastrointestinal abnormalities
7. Severe clinical condition / disorders which the Investigator considers a contraindication to study participation, including the presence of at least 3 out of 4 of the following symptoms:

   1. necessity of mechanical ventilation and FiO2 more than 0.6 elevation to maintain blood oxygen saturation within 88-93%,
   2. metabolic acidosis, pH less than 7.20 and BE more than (-10),
   3. necessity of vasopressor (antihypotensive) agents to maintain proper arterial blood pressure,
   4. signs of damage to at least one vital organ (liver, kidneys, gastrointestinal tract, adrenal glands).
8. Administration of other probiotic preparations
9. Enrolment in any other clinical trial throughout the study period
10. Lack of parent-legal guardian informed consent

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 182 (Actual)
Dates: Start 2012-04; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal tract colonisation | Assesed on days 1, 7, 14, 21, 28, 35, 42 and 49 (assesed weekly within eight weeks)
  Bacteriological tests involved quantitative and qualitative assessment of neonatal gut flora during clinical follow-up. Bacterial populations of Lactobacillus and Bifidobacterium as well as pathogenic bacteria were assesed.
  Stool samples were collected at 7-day intervals (±2 days) in the period of investigational product intake, and on Day 7 (±2 days) after the last dose of the investigational product.
Feeding intolerance episodes (including: gastric residuals, vomiting, regurgitation of food, abdominal distension, abdominal rigidity, gut motility disorders) | Assesed on a daily basis (from 1 to 42 and on day 49)
  Clinical parameters were evaluated throughout the period of care according to standard neonatal care procedures.
Incidence and type of adverse events and serious adverse events with special regard to sepsis caused by bacteria contained in investigational product. | Assesed on a daily basis (from 1 to 42 and on day 49)
  Safety was evaluated by determining whether investigational product in VLBW preterm neonates increases AE/SAE incidence and influences the type of adverse events and serious adverse events as compared to placebo with special regard to sepsis caused by bacteria contained in investigational product .

SECONDARY OUTCOMES:
Late onset sepsis caused by Gram positive or Gram negative bacteria | Assesed on a daily basis (from 1 to 42 and on day 49)
  Sepsis was confirmed by positive blood cultures. Clinical parameters were evaluated throughout the period of care according to standard neonatal care procedures.
Gastrointestinal perforation | Assesed on a daily basis (from 1 to 42 and on day 49)
  Clinical parameters were evaluated throughout the period of care according to standard neonatal care procedures.
Duration of total parenteral nutrition (days) | Assesed on a daily basis (from 1 to 42 and on day 49)
  Duration of total parenteral nutrition (hyperalimentation) was evaluated until full enteral nutrition is restored.
Duration (days) of absence of enteral nutrition due to gastrointestinal disorders | Assesed on a daily basis (from 1 to 42 and on day 49)
  Clinical parameters were evaluated throughout the period of care according to standard neonatal care procedures.
Duration (days) of absence of enteral nutrition for reasons other than gastrointestinal disorders | Assesed on a daily basis (from 1 to 42 and on day 49)
  Clinical parameters were evaluated throughout the period of care according to standard neonatal care procedures.
Weight, length and head circumference | Weight was measured once daily, head circumference was measured once a week, and body length was measured on Day 1 and on Day 7 (±2 days) from the last dose (or until the patient was discharged or withdrawn from the study)
  Weight, length and head circumference were evaluated throughout the period of care according to standard neonatal care procedures.
NEC - intensity and severity | Assesed on a daily basis (from 1 to 42 and on day 49)
  Severity of neonatal necrotizing enterocolitis was determined according Bell's criteria. Clinical parameters were evaluated throughout the period of care according to standard neonatal care procedures.
Mortality rate, with a focus on deaths attributed to NEC and sepsis | Assesed on a daily basis (from 1 to 42 and on day 49)
  Clinical parameters were evaluated throughout the period of care according to standard neonatal care procedures.
Duration of hospitalization (days) (until discharge) | Assesed on a daily basis (from 1 to 42 and on day 49)
  Duration of hospitalization was investigated from the date of patient enrolment until discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Ryszard Lauterbach, Prof., MD, Principal Investigator — Jagiellonian University Medical College, Department of Neonatology, Kopernika 23 St., 31-501 Krakow, Poland; Aleksandra M Cichonska, PhD, Study Director — IBSS Biomed S.A.